CLINICAL TRIAL: NCT01967667
Title: Biological Evaluation of Dietary Supplement Liposomal Glutathione
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HP-00056458
Record Dates: First submitted 2013-10-17; First posted 2013-10-23 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — glutathione pegylated liposomal doxorubicin; Glutathione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal glutathione (Experimental): dose steps
  Interventions: Dietary Supplement: Liposomal glutathione
- Placebo (Placebo Comparator): dose steps
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Liposomal glutathione — Escalating dose steps
  Other Names: ReadiSorb glutathione
  Arms: Liposomal glutathione
Dietary Supplement: Placebo — escalating dose steps
  Other Names: Readisorb solution without glutathione
  Arms: Placebo

SUMMARY:
Low levels of antioxidant molecules such as glutathione have been found in people with a diagnosis of schizophrenia. However, oral glutathione is not well absorbed because the compound is mostly broken down in the gastrointestinal system. Liposomes are tiny droplets of oil particles that encapsulate and protect the glutathione. In this study we will evaluate a liposomal formulation of glutathione for tolerability and to examine if this formulation serves the function of increasing glutathione in the brain and body.

DETAILED DESCRIPTION:
Additional information about this dietary supplement:

* Glutathione is an antioxidant naturally produced in our body. Glutathione protects the brain and other organs from oxidative stress.
* Low glutathione is associated with high oxidative stress, which has been linked to aging and many illnesses. Schizophrenia is a mental illness that doctors still do not fully understand. Individuals with schizophrenia often have low levels of glutathione.
* Glutathione can be supplied through dietary supplement. However, if taken plainly, it easily breaks down in our gut.
* Scientists have now found a way to wrap glutathione in tiny drops of oil particles called liposomes. That way, the gut cannot break it down so it is absorbed into our body. Once inside the body, our cells can take in the liposomes and use the glutathione to reduce oxidative stress.
* Liposome-wrapped glutathione is not a drug or medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-60
* DSM diagnosis of schizophrenia spectrum disorder, including schizophrenia, schizoaffective disorder, and schizophreniform disorder
* Ability to give written informed consent (Evaluation to Sign Consent score 10 or greater)
* Clinically stable with no change in antipsychotic medications nor significant increase of daily dose for 2 weeks prior to enrollment
* Low baseline blood glutathione level (GSH < 890 umol/l)

Exclusion Criteria:

* History of major medical illness including, but not limited to, history of heart attack, stroke, TIA (transient ischemic attack)
* History of organic brain disorders that may affect neurophysiological measurements, including seizure disorder, brain tumor, head injury with evidence of significant cognitive deterioration
* DSM diagnosis of substance dependence within 6 months except nicotine and marijuana, or substance abuse in past month
* Uncontrolled blood pressure (persistent systolic above 165 or diastolic above 100)
* On medication containing cholesterol absorption inhibitor such as ezetimibe (Brand names Zetia, Ezetrol, Vytorin, and Inegy)
* Women who have positive urine pregnancy tests
* Women who plan to become pregnant, or are breastfeeding
* Unable to undergo MRI scanning due to metallic devices or objects or claustrophobia
* Already taking dietary antioxidant supplements such as n-acetylcysteine or fish oil on regular basis (more than twice a week) in the last 3 months
* History of allergy to soy or soy products
* Hyperlipidemia (baseline LDL > 1.5 x upper limit of normal)
* Liver impairment (baseline AST or ALT > 2.0 x upper limit of normal)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Glutathione levels | Baseline and 3 weeks
  Change of glutathione levels from baseline to following 3 weeks of treatment.

SECONDARY OUTCOMES:
oxidative stress biomarker | baseline and 3 weeks
  blood levels of lipid peroxidation
inflammatory marker | baseline and 3 weeks
  Blood levels of cytokines as biomarkers of inflammation

OTHER OUTCOMES:
BPRS | Baseline and 3 weeks
  Change in brief psychiatric rating scale scores from baseline to end of treatment phase and end of placebo phase.
Adverse events | Baseline and 3 weeks
  side-effects checklist

CONTACTS AND LOCATIONS:
Overall Officials: L. Elliot Hong, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No